CLINICAL TRIAL: NCT02996071
Title: May Preoperative Waist to Height Ratio Predict Postoperative Weight Loss in Bariatric Patients?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016_10/16
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low waist to height ratio (Active Comparator): laparoscopic sleeve gastrectomy
  Interventions: Procedure: laparoscopic sleeve gastrectomy
- high waist to height ratio (Active Comparator): laparoscopic sleeve gastrectomy
  Interventions: Procedure: laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy — a sleeve gastrectomy operation that is performed laparoscopically.

SUMMARY:
Bariatric surgery is an effective method for treatment of obesity. Sleeve gastrectomy is one of surgical methods and became popular in recent years. Weight loss rates after bariatric surgery differs among patients. The exact reason of this difference stays unclear. age, nationality, difference between body composition and type of surgery may be in concern. waist to height ratio has become popular recent years as an indicator of cardiomethabolic status. in this study, investigation of the effect of waist to height ratio differences of patients on weight loss following laparoscopic sleeve gastrectomy as a bariatric surgery.

DETAILED DESCRIPTION:
Waist to height raito is the major determinator of patients and will be noted in every patient who will fulfil the eligibility criteras defined below and undergo laparoscopic sleeve gastrectomy. demographic data, BMI, body lipid composition, lean body weight also will be noted. all patients will undergo standardized laparoscopic sleeve gastrectomy operation. patients will be follow up during first, third, sixth and one year periods. all parameters noted preoperatively will be measured and noted again. possible statistical difference will be calculated statistically and a cut off value will be seeked.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* BMI>40 kg/m2
* Sleeve gastrectomy operation planned patients

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* osteoarticular pathology that may restrict postoperative regular physical activity.
* apparent mental or psychological disorder that may affect postoperative recommendations
* refusal of informed consent for this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
weight loss rates | 6 months

SECONDARY OUTCOMES:
overall complications | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin K Bektasoglu, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided